CLINICAL TRIAL: NCT02259686
Title: Cardiovascular Effects of Apelin In Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Apelin2014
Record Dates: First submitted 2014-10-01; First posted 2014-10-08 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Apelin; volunteers
MeSH Terms: interventions — Apelin; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protocol 1. Apelin 1mg doses (Experimental): 5 Healthy volunteers
  Interventions: Drug: Apelin 1mg subcutaneous; Drug: Apelin 1mg intravenous
- Protocol 2. Apelin 5mg doses (Experimental): 5 Healthy volunteers
  Interventions: Drug: Apelin 5mg subcutaneous; Drug: Apelin 5mg intravenous
- Protocol 3. Apelin 10mg single dose (Experimental): 5 Healthy volunteers
  Interventions: Drug: Apelin 10 mg subcutaneous

INTERVENTIONS:
Drug: Apelin 1mg subcutaneous — single subcutaneous injection of Apelin 1mg subcutaneous
  Other Names: 1mg Sc
  Arms: Protocol 1. Apelin 1mg doses
Drug: Apelin 1mg intravenous — 15 minute intravenous bolus of Apelin 1mg intravenous
  Other Names: 1mg iv
  Arms: Protocol 1. Apelin 1mg doses
Drug: Apelin 5mg subcutaneous — single subcutaneous injection of Apelin 5mg subcutaneous
  Other Names: 5mg Sc
  Arms: Protocol 2. Apelin 5mg doses
Drug: Apelin 5mg intravenous — 15 minute intravenous infusion of Apelin 5mg intravenous
  Other Names: 5mg iv
  Arms: Protocol 2. Apelin 5mg doses
Drug: Apelin 10 mg subcutaneous — 24 hour continuous subcutaneous infusion of Apelin 10 mg subcutaneous
  Other Names: 10mg sc
  Arms: Protocol 3. Apelin 10mg single dose

SUMMARY:
Apelin is an endogenous peptide with physiological actions in the cardiovascular system. Apelin can modulate vasomotor tone and is a potent endogenous inotrope. In a series of clinical studies, we have shown that apelin causes peripheral and coronary vasodilatation and increased cardiac contractility. We wish to study and compare the cardiovascular effects of subcutaneous versus intravenous apelin. We specifically wish to determine how different methods of apelin administration affect cardiac output and peripheral vascular resistance in healthy volunteers

DETAILED DESCRIPTION:
Study Protocols Groups of 5 subjects will be assigned to receive one of three protocols.

Protocol 1:

Five healthy volunteers will be asked to attend the clinical research facility on a total of 4 occasions as per the protocol below.

Visits 1 and 2 will occur over two consecutive days. Participants will attend at 07.30 and be given a light breakfast. An intravenous sampling cannula will be inserted into the antecubital vein of one arm. Blood samples (5 mL) will be taken immediately prior to subcutaneous injection (t=0; 08.00) of 1 mg (Pyr1)apelin-13 and at 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 600 min after injection. Subjects will then be discharged from the facility and reattend the following day at 08.00 for a single venous sample. Approximately 85 mL of blood will be sampled in total over this time.

Visits 3 and 4 will also occur over two consecutive days, at least one week after visit 2. Subjects will attend at 07.30 and be given a light breakfast. An intravenous sampling cannula will be inserted into the antecubital vein of one arm. Blood samples (5 mL) will be taken immediately prior to an intravenous bolus infusion (t=0; 08.00) of 1 mg (Pyr1)apelin-13 over 15 min and at 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 600 min after injection. Subjects will then be discharged from the facility and reattend the following day at 08.00 for a single venous sample.

Protocol 2:

Five healthy volunteers will be asked to attend the clinical research facility on a total of 4 occasions as per the protocol below.

Visits 1 and 2 will occur over two consecutive days. Participants will attend at 07.30 and be given a light breakfast. An intravenous sampling cannula will be inserted into the antecubital vein of one arm. Blood samples (5 mL) will be taken immediately prior to subcutaneous injection (t=0; 08.00) of 5 mg (Pyr1)apelin-13 and at 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 600 min after injection. Subjects will then be discharged from the facility and reattend the following day at 08.00 for a single venous sample. Approximately 85 mL of blood will be sampled in total over this time.

Visits 3 and 4 will also occur over two consecutive days, at least one week after visit 2. Subjects will attend at 07.30 and be given a light breakfast. An intravenous sampling cannula will be inserted into the antecubital vein of one arm. Blood samples (5 mL) will be taken immediately prior to an intravenous bolus infusion (t=0; 08.00) of 5 mg (Pyr1)apelin-13 over 15 min and at 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 600 min after injection. Subjects will then be discharged from the facility and reattend the following day at 08.00 for a single venous sample.

Protocol 3:

Five healthy volunteers will be asked to attend the clinical research facility for 2 consecutive days. Subjects will attend at 07.30 and be given a light breakfast. An intravenous sampling cannula will be inserted into the antecubital vein of one arm. Blood samples (5 mL) will be taken immediately prior to commencing a 24-h subcutaneous infusion of (t=0; 08.00) of 10 mg (Pyr1)apelin-13 dissolved in 10 mL water for injection. Further venous sampling will take place at 5, 10, 15, 20, 25, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 600 min after injection. Subjects will then be discharged from the facility and reattend the following day at 08.00 for a single venous sample.

Measurements

Thoracic Bioimpedance Cardiography By virtue of changes in transthoracic electrical impedance during cardiac ejection, thoracic bioimpedance cardiography allows the non-invasive assessment of cardiac stroke volume and the calculation of cardiac output and cardiac index. After skin preparation, four pairs of low-contact impedance 'sensing' and 'current injecting' electrodes will be attached to the patient and connected to an impedance cardiograph. This technique has been applied widely and compares favourably with both invasive and other non-invasive (echocardiographic) measures of cardiac output. These variables will therefore be recorded at regular intervals throughout the study in all 3 protocols. Heart rate and blood pressure will also be monitored at regular intervals throughout each study using a semi-automated oscillometric sphygmomanometer (Omron HEM-705CP, Omron, Matsusaka, Japan). Mean arterial pressure (MAP) will be calculated as diastolic blood pressure plus a third of the pulse pressure.

Assays Blood samples (5 mL) will be collected before and at the end of each drug infusion into ethylene diamine tetraacetic acid (EDTA), centrifuged and plasma frozen in three 1-mL aliquots to be stored at -80 °C until assay. Plasma concentrations of apelin will be measured by collaborators at Bristol Myers Squibb, Princeton, USA.

Methods of Statistical Analysis

Outcome data will be analysed where appropriate, by analysis of variance (ANOVA) with repeated measures, regression analysis, and paired and unpaired Student's t-test. Statistical significance will be taken at the 5% level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females >18 years old
* Willing and able to complete an informed consent form

Exclusion Criteria:

* Unable to give informed consent
* Pregnant or lactating at screening
* Use of any investigation product or device within 30 days prior to study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output between different methods of apelin administration. | 10 hours
  Difference in cardiac output between different treatment arms. This will be assessed by recording cardiac index in L/min/m2 and Stroke volume index mL/min/m2
Change in blood pressure between different methods of apelin administration. | 10 hours
  Difference in blood pressure between different treatment arms assessed by measuring mean blood pressure in mmHg. Mean arterial pressure (MAP) will be calculated as diastolic blood pressure plus a third of the pulse pressure

SECONDARY OUTCOMES:
Change in apelin concentrations between the different methods of administration | 24 hours
  Difference in temporal profile of apelin concentrations produced by different methods of apelin administration

CONTACTS AND LOCATIONS:
Overall Officials: David Newby, Principal Investigator — British Heart Foundation
Locations (2):
- United Kingdom (2):
  - Clinical Research Facility University of Edinburgh, Edinburgh
  - Wellcome Trust Clinical Research Facility. Western General Hospital, Edinburgh